CLINICAL TRIAL: NCT02063685
Title: A Multicenter, Phase III, Randomized Study to Evaluate the Efficacy of Response-adapted Strategy to Define Maintenance After Standard Chemoimmunotherapy in Patients With Advanced-stage Follicular Lymphoma.
Brief Title: Study to Evaluate the Efficacy of Response-adapted Strategy in Follicular Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_FOLL12
Record Dates: First submitted 2013-11-21; First posted 2014-02-14 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Follicular Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Bendamustine Hydrochloride; Observation; ibritumomab tiuxetan; Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- GROUP 1 - STANDARD (Other): R-CHOP or R-bendamustine + Standard Maintenance
  Interventions: Drug: R-CHOP or R-bendamustine; Drug: Standard Maintenance
- GROUP 2 (Experimental): FDG-PET POSITIVE (score 4-5) patients (High risk) R-CHOP or R-bendamustine + Ibritumomab Tiuxetan + Maintenance
  Interventions: Drug: R-CHOP or R-bendamustine; Drug: Ibritumomab Tiuxetan + Maintenance
- GROUP 1a (Experimental): FDG-PET NEGATIVE (score 1-3) AND MRD NEGATIVE R-CHOP or R-bendamustine + Observation
  Interventions: Drug: R-CHOP or R-bendamustine; Drug: Observation
- GROUP 1b (Experimental): FDG-PET NEGATIVE (score 1-3) AND MRD POSITIVE R-CHOP or R-bendamustine + Maintenance weekly x4
  Interventions: Drug: R-CHOP or R-bendamustine; Drug: Maintenance weekly x4

INTERVENTIONS:
Drug: R-CHOP or R-bendamustine — As induction therapy all patients will receive 6 courses of:
  Rituximab: 375 mg/m² day 1 iv Cyclophosphamide: 750 mg/m² day 1 iv Doxorubicin: 50 mg/m² day 1 iv Vincristine: 1.4 mg/m² day 1 iv (max dose 2mg) Prednisone: 100 mg day 1-5 os To allow administration of all drugs on the same day, Rituximab rapid infusion is permitted starting from cycle 2. Cycles are to be repeated every 21 days.
  or 6 courses of:
  Rituximab: 375 mg/m² day 1 iv Bendamustine: 90 mg/m² day 1 and 2 iv. To allow administration of all drugs on the same day, Rituximab rapid infusion is permitted starting from cycle 2. Cycles are to be repeated every 28 days.
  Other Names: Rituximab; Cyclophosphamide,; Hydroxydaunorubicin; Oncovin; Prednisone; Bendamustine
Drug: Observation — not maintenance therapy and followed-up with MRD monitoring.
  Arms: GROUP 1a
Drug: Maintenance weekly x4 — Four weekly doses of Rituximab (375 mg/m²). Rituximab could be repeated for MRD positive for a maximum of three courses
  Other Names: Rituximab
  Arms: GROUP 1b
Drug: Ibritumomab Tiuxetan + Maintenance — single dose of (90)Y Ibritumomab Tiuxetan (0.4 mCi/kg). Following RIT patients will continue maintenance with Rituximab (375 mg/m² every 2 months) for a total of 11 infusions.
  Other Names: Ibritumomab Tiuxetan
  Arms: GROUP 2
Drug: Standard Maintenance — Rituximab 375 mg/m² every 2 months for 2 years. Maintenance will have to be started no more than 12 weeks after the last induction chemoimmunotherapy infusion.
  Other Names: Rituximab
  Arms: GROUP 1 - STANDARD

SUMMARY:
Recently, the availability of R has substantially changed therapeutic approach to FL patients, since its combination with chemotherapy has improved response rates, progression free survival (PFS) and overall survival (OS). Based on the results of recently completed randomized studies the standard treatment for patients with FL should consist of an initial therapy with R-CHOP combination followed by two-year maintenance with R. Although results of randomized trials confirmed that this approach results in an improved patients' outcome and made a step forward in the management of patients with FL, one important question that can be raised is if this approach is really needed for all patients with FL or if some of them could benefit from a reduced intensity treatment achieving the same results in terms of outcome and survival . This question is of particular interest for newly diagnosed patients for whom maintenance does not affect OS.

More recent data demonstrated that the outcome of patients with FL can be further predicted by evaluating the quality of response to therapy studying minimal residual disease (MRD). This project addresses the objective of evaluating if combining clinical response assessed on FDG-PET scan and molecular response measured through MRD detection could permit to single out groups of patients at different risk of progression and to consequently modulate maintenance therapies, with the aim to provide clinicians a more rational use of the available diagnostic and therapeutic resources.

DETAILED DESCRIPTION:
This is a multicenter, randomized, phase III, superiority study comparing standard vs response driven approach to maintenance. Adult patients (age ≥ 18 years) with naïve, untreated follicular lymphoma, stage II-IV, Follicular Lymphoma International Prognostic Index 2 (FLIPI2) >0 requiring a therapeutic intervention will be recruited and randomly assigned in a 1:1 ratio to either standard or experimental arm.

All patients will receive the same induction therapy with 6 cycles of R-CHOP or R-bendamustine and 2 additional doses of Rituximab.

At baseline patients will be assessed for molecular status and staged by means of CT scan. A baselineFluorine-18-Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) scan should also be performed.

At the end of chemoimmunotherapy all patients will be assessed for disease response by common clinical and laboratory examination, CT scan and FDG-PET. An intermediate assessment of response with CT scan and FDG-PET (optional) will also be performed after the first four courses of R-chemoimmunotherapy.

At the end of induction therapy the status of minimal residual disease will be also evaluated.

After induction treatment all responding patients in the standard arm will receive standard maintenance therapy with Rituximab (every 2 months for 2 years), while patients in the experimental arm will be subdivided into two risk groups and assigned to different post induction treatments based on FDG-PET and MRD results. In both arms, patients with stable or progressive disease (PET positive and less than PR on CT scan) will be addressed to salvage treatment chosen at physician discretion.

In the experimental arm, risk group allocation will be performed primarily on the basis of FDG-PET results:

* Group 1 (low risk): negative FDG-PET
* Group 2 (high risk): positive FDG-PET

Patients at low risk (FDG-PET negative) will received maintenance therapy according to their MRD status,particularly:

* Group 1a (MRD negative): observation
* Group 1b (MRD positive): pre-emptive Rituximab therapy

Patient at high risk (FDG-PET positive) will receive maintenance regardless of their MRD status:

· Group 2: intensified maintenance ((90)Y Ibritumomab Tiuxetan + Rituximab maintenance )

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of B-Cell CD20+ Follicular Lymphoma (FL), grade I, II, IIIa according to the WHO 2008 classification
* ECOG performance status 0-2
* Age ≥ 18 years
* Ann Arbor stage II-IV
* FLIPI2>0
* Presence of evaluable/measurable disease after diagnostic biopsy
* At least one of the following criteria for defining active disease:

  * systemic symptoms
  * cytopenia due to bone marrow involvement
  * LDH> upper normal value
  * any nodal or extranodal tumor mass with a diameter >7cm
  * involvement of ≥ 3 nodal sites, each with a diameter of ≥ 3cm
  * extranodal disease
  * rapidly progressive disease
* Life expectancy > 6 months
* Left ventricular ejection fraction (LVEF) ³ 50%
* Serum negativity for HIV
* Serum negativity for HBsAg; HBcAb positive but HBV-DNA negative patients are allowed with mandatory Lamivudine prophylaxis.
* Serum negativity for HCV, except for those patients without signs of active viral replication assessed by HCV-RNA copies
* Serum creatinine < 2mg/dl , serum bilirubin < 1.5mg/dl, aspartate amino-transferase (AST/GOT) £ 2.5xUNV, alanine amino-transferase (ALT/GPT) £ 2.5xUNV, and alkaline phosphatase £ 4 times the upper limit of normal (unless the increase is attributed directly to the presence of tumour by the Investigator)
* Patients with no previous treatment for the lymphoma with the exception of locoregional radiotherapy (IFRT)
* Adequate measure adoption to avoid pregnancy
* Written informed consent given at time of registration
* Patient must be accessible for treatment and follow up.

Exclusion Criteria:

* Histological diagnosis of :

  * any lymphoma other than follicular lymphoma and all CD20 negative B-cell lymphomas
  * grade III b follicular lymphoma
  * evidence of transformation to high grade lymphoma
* Ann Arbor stage I
* Suspect or clinical evidence of CNS involvement by lymphoma
* History of other malignancies within 5 years prior to study entry except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer, low grade, early stage localized prostate cancer treated surgically with curative intent, good prognosis DCIS of the breast treated with lumpectomy alone with curative intent
* Evidence of any severe active acute or chronic infection
* Concurrent co-morbid medical condition which might exclude administration of full dose chemotherapy
* Severe chronic obstructive pulmonary disease with hypoxemia
* Severe diabetes mellitus difficult to control with adequate insulin therapy
* Myocardial infarction within 6 months before study entry
* Clinically significant secondary cardiovascular disease e.g. uncontrolled hypertension, (resting diastolic blood pressure >115 mmHg), uncontrolled multifocal cardiac arrhythmias, symptomatic angina pectoris or congestive cardiac failure NYHA class III-IV
* HbsAg-positive, HIV-positive, or HCVAb-positive patients
* Known hypersensitivity or anaphylactic reactions to murine antibodies or proteins
* Any other co-existing medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent
* Follicular lymphoma, showing a negative baseline PET scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 807 (Actual)
Dates: Start 2012-07; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
PFS | 12/31/2019
  To evaluate whether a FDG-PET and MRD response-based maintenance therapy is more effective in terms of Progression-Free Survival (PFS) than a standard maintenance therapy with Rituximab in patients with untreated, advanced, follicular lymphoma. Progression Free Survival (PFS) PFS will be measured from the date of randomization to the date of documented first occurrence of disease progression or relapse or to the date of death from any cause. Responding patients and patients who are lost to follow up will be censored at their last assessment date.

SECONDARY OUTCOMES:
CRR | 12/31/2019
  Complete Response Rate (CRR) is defined as the number of CR after the completion of the study treatment. Patients without a response assessment (due to any reasons) will be considered as non-responders.
ORR | 12/31/2019
  Overall Response Rate (ORR) after the completion of the treatment, defined as the sum of Complete Response and Partial Response. Patients without a response assessment (due to any reasons) will be considered as non-responders.
DR | 12/31/2019
  Duration of Response (DR) is from the time when criteria for response (ie, CR or PR) are met, to the first documentation of relapse or progression.
EFS | 12/31/2019
  Event Free Survival (EFS) is measured from the time from study entry to any treatment failure including disease progression, or discontinuation of treatment for any reason (eg, disease progression, toxicity, patient preference, initiation of new treatment without documented progression, or death).
OS | 12/31/2019
  Overall survival (OS) is defined as the time from the first day of study treatment until the date of death irrespective of cause. Patients who have not died at the time of end of the whole study , and patients who are lost to follow up , will be censored at the date of the last contact.
Molecular response analysis | 12/31/2019
  * Rate of molecular remission will be defined as the proportion of patients polymerase chain reaction (PCR) negative for Bcl2/IgH at different time-points including those achieving continuous MR in two or more consecutive time-points. Patients without a response assessment (due to any reasons) will be excluded from the analysis.
  * Rate of conversion will be defined as the proportion of patients from baseline PCR-positivity to PCR-negativity. Patients without a response assessment (due to any reasons) will be excluded from the analysis.
  * Rate of molecular relapse will be defined as the proportion of patients from PCR-negativity to PCR-positivity. Patients without a response assessment (due to any reasons) will be excluded from the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Donato Mannina, MD, Principal Investigator — Hematology, Azienda Ospedali Riuniti Papardo-Piemonte, Messina, Italy.; Massimo Federico, MD, Principal Investigator — Department of Diagnostic Medicine, Clinical Medicine and Public Health, University of Modena and Reggio Emilia, Modena , Italy
Locations (48):
- Italy (48):
  - Irst - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori - Sede Di Meldola (Fc), Meldola, Forlì Cesena
  - ASUR 8, Civitanova Marche, Macerata
  - Irccs Istituto Clinico Humanitas, Rozzano, Milano
  - Fondazione IRCCS Milano INT, Milan, MI
  - Azienda Ospedaliera S. Gerardo Di Monza, Monza, Monza Brianza
  - Irccs Centro Di Riferimento Oncologico Di Basilicata (Crob), Rionero in Vulture, Potenza
  - P.O. Umberto I, Nocera Inferiore, Salerno
  - Fondazione Del Piemonte Per L'Oncologia Ircc Di Candiolo, Candiolo, Torino
  - A.O. S. Maria di Terni, Terni, TR
  - Ospedale Civile Ss. Antonio E Biagio Di Alessandria - Alessandria (Al), Alessandria
  - A.O. Universitaria Ospedali Riuniti - Ospedale Umberto I Di Ancona _, Ancona
  - A.O. Universitaria Ospedale Consorziale Policlinico Di Bari, Bari
  - A.O. Ospedale Degli Infermi, Biella
  - A.O. Universitaria Policlinico S.Orsola-Malpighi Di Bologna, Bologna
  - Pres.Ospedal.Spedali Civili Brescia, Brescia
  - Stabilimento "Perrino" - Brindisi -, Brindisi
  - Ospedale Armando Businco - Cagliari, Cagliari
  - A.O. Universitaria Ospedale Vittorio Emanuele Di Catania, Catania
  - Azienda Ospedaliera S. Croce E Carle Di Cuneo, Cuneo
  - A.O. Universitaria Careggi Di Firenze, Florence
  - A.O. Universitaria S. Martino Di Genova, Genova
  - Ematologia Ospedale Vito Fazzi, Lecce
  - Presidio Ospedaliero - Matera -, Matera
  - Azienda Ospedaliera Papardo, Messina
  - Irccs Ospedale Maggiore Policlinico Di Milano, Milan
  - Ospedale Ca' Granda-Niguarda, Milan
  - A.O. Universitaria Policlinico Di Modena, Modena
  - Irccs Istituto Nazionale Tumori Fondazione Pascale, Napoli
  - A.O. Universitaria Maggiore Della Carita' Di Novara, Novara
  - Ospedale San Francesco, Nuoro
  - A.O. Universitaria Policlinico Giaccone Di Palermo, Palermo
  - A.O. "V. Cervello", Palermo
  - A O Universitaria di Parma, Parma
  - IRCCS Policlinico S. Matteo, Pavia
  - Azienda Ospedaliera Di Perugia - Ospedale S. Maria Della Misericordia -, Perugia
  - Ospedale Civile Spirito Santo, Pescara
  - Ausl Di Piacenza, Piacenza
  - A.O. Universitaria Pisana, Pisa
  - Ospedale Bianchi - Melacrino - Morelli, Reggio Calabria
  - Ausl Di Rimini, Rimini
  - Universita' Degli Studi Di Roma 'La Sapienza', Roma
  - Casa sollievo della Sofferenza, San Giovanni Rotondo
  - A.O. Universitaria Senese, Siena
  - A.O. Universitaria S. Giovanni Battista-Molinette Di Torino, Torino
  - Ospedale Ca Foncello, Treviso
  - A.O.Cardinale Panico Ematologia e centro trapianti, Tricase (LE)
  - A.O. Universitaria S. Maria Della Misericordia Di Udine, Udine
  - Ospedale Di Circolo E Fondazione Macchi, Varese

REFERENCES:
- [Derived] Durmo R, Chauvie S, Fallanca F, Bergesio F, Pinto A, Del Giudice I, Coscia M, Corradini P, Angelucci E, Tosi P, Freilone R, Ballerini F, Bari A, Pastore D, Zinzani PL, Bolis S, Flenghi L, Liso A, Olivieri J, Marcheselli L, Merli M, Versari A, Guerra L, Luminari S. Prognostic role of interim PET in follicular lymphoma: a post hoc study of FOLL12 trial by Fondazione Italiana Linfomi. Blood Adv. 2025 Jun 24;9(12):2927-2934. doi: 10.1182/bloodadvances.2024014790. PMID 40106688
- [Derived] Luminari S, Manni M, Galimberti S, Versari A, Tucci A, Boccomini C, Farina L, Olivieri J, Marcheselli L, Guerra L, Ferrero S, Arcaini L, Cavallo F, Kovalchuk S, Skrypets T, Del Giudice I, Chauvie S, Patti C, Stelitano C, Ricci F, Pinto A, Margiotta Casaluci G, Zilioli VR, Merli A, Ladetto M, Bolis S, Pavone V, Chiarenza A, Arcari A, Anastasia A, Dondi A, Mannina D, Federico M; Fondazione Italiana Linfomi. Response-Adapted Postinduction Strategy in Patients With Advanced-Stage Follicular Lymphoma: The FOLL12 Study. J Clin Oncol. 2022 Mar 1;40(7):729-739. doi: 10.1200/JCO.21.01234. Epub 2021 Oct 28. PMID 34709880